CLINICAL TRIAL: NCT04546893
Title: Safety and Efficacy Study of SL1904B CAR-T Cells for Relapsed or Refractory B-Cell Acute Lymphocyte Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other); Beijing Lu Daopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1904B for B-ALL
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: B-ALL
Keywords: B-ALL, CD19 CAR-T

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1904B CAR-T (Experimental): Patients will be treated with CD19 CAR-T cells
  Interventions: Biological: CD19 CAR-T

INTERVENTIONS:
Biological: CD19 CAR-T — Biological: CD19 CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis;

SUMMARY:
This is an open, single-arm, clinical study to evaluate efficacy and safety of anti CD19 CAR-T cell in the treatment of recurrent or refractory B-ALL

DETAILED DESCRIPTION:
The CARs consist of an anti-CD19 single-chain variable fragment（scFv） that was derived from the FMC63 mouse hybridoma, a portion of the human CD137（4-1BB） molecule, and the intracellular component of the human CD3ζ molecule. Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

The Main research objectives:

To evaluate the safety and efficacy of 1904B in patients with recurrent or refractory B-ALL

The Secondary research objectives:

To investigate the cytokinetic characteristics of 1904B in patients with recurrent or refractory B-ALL

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent and be willing and able to comply with the visit, treatment regimen, laboratory examination and other requirements of the study as stipulated in the trial flow chart;
2. A definite diagnosis of B-cell Lymphocyte Leukemia, which meets any of the following criteria: Relapsed : a) relapsed within 12 months after first remission;Refractory: a) no remission after six weeks of induction therapy or no remission after two courses of induction therapy; b) relapsedafter CR for 2 or more times; c) The first relapse after chemotherapy and no remission after at least one salvage treatment; c) relapsed after hematopoietic stem cell transplantation;
3. ECOG Scores: 0~2
4. CD19 positivewere detected by immunohistochemistry or flow cytometry;
5. Estimated survival time>3 months;
6. Peripheral blood mononuclear immune cells must be collected at least 2 weeks after the last radiotherapy or systemic treatment.

Exclusion Criteria:

1. Serious cardiac insufficiency；
2. Has a history of severe pulmonary function damaging;
3. With other tumors which is/are in advanced malignant and has/have systemic metastasis;
4. Severe or persistent infection that cannot be effectively controlled；
5. Merging severe autoimmune diseases or immunodeficiency disease;
6. Patients with active hepatitis B or hepatitis C([HBVDNA+]or [HCVRNA+]);
7. Patients with HIV infection or syphilis infection;
8. Has a history of serious allergies on Biological products (including antibiotics);
9. Being pregnant and lactating or having pregnancy within 12 months;
10. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after SL1904B infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  Remission Rate including complete remission(CR)、CR with incomplete blood count recovery(CRi)、No remission(NR)

SECONDARY OUTCOMES:
Efficacy:duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD19 CAR- T cells in the genomes of PBMC by qPCR method and percentage of CD19 CAR- T cells measured by flow cytometry method
Cytokine release | First month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (2):
- China (2):
  - Hebei yanda Ludaopei Hospital, Hebei, Sanhe
  - BeiJing Ludaopei Hospital, Beijing, Yizhuang